CLINICAL TRIAL: NCT01206270
Title: Androgen Treatment in Leydig Cell Proliferation
Brief Title: Androgen for Leydig Cell Proliferation
Acronym: ALCeP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, Professor of Endocrinology, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 160/10
Record Dates: First submitted 2010-09-09; First posted 2010-09-21 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Klinefelter Syndrome; Hypergonadotropic Hypogonadism; Hypergonadotropic Azospermia; Hypergonadotropic Cryptozoospermia
Keywords: Klinefelter; Leydig; Testicular Tumor; LH; Infertility
MeSH Terms: conditions — Klinefelter Syndrome; Hypogonadism; Testicular Neoplasms; Infertility | interventions — testosterone undecanoate; Castor Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone (Experimental): Testosterone undecanoate 1000mg injection at baseline (0-week), 6-week, 18-week, 30-week
  Interventions: Drug: Testosterone undecanoate
- Placebo (Placebo Comparator): Injection 4 ml of castor oil at baseline (week-0), week-6, week-18, week-30
  Interventions: Drug: Castor Oil

INTERVENTIONS:
Drug: Testosterone undecanoate — Testosterone undecanoate 1000mg (in 4 ml of castor oil injections) at baseline (0-week), 6-week, 18-week, 30-week
  Other Names: Nebido
  Arms: Testosterone
Drug: Castor Oil — 4 ml of Castor Oil injected at baseline (0-week), 6-week, 18-week, 30-week.
  Arms: Placebo

SUMMARY:
Patients with infertility often presents alterations at ultrasonographic examination of the testis. These alterations include a much higher incidence of small, multiple, non-palpable hypoechoic micro-nodules that can show internal vascularization. This finding often create alarm and anxiety, because it has to be placed in a differential diagnosis versus low-stage malignant germ cell tumors. Nevertheless, explorative surgery reveal that a consistent number of these lesion are benign, due to Leydig cell hyperplasia or Leydig cell tumours. The purpose of this study is to evaluate the effects of androgen therapy on the size and number of non-palpable hypoechoic micro-nodules in patients with elevated gonadotropin levels.

DETAILED DESCRIPTION:
Patients with the testicular dysgenesis syndrome, that comprises a variable spectrum of clinical manifestations, such as infertility, cryptorchidism, hypospadias, impaired spermatogenesis and testicular germ cell neoplasms, often develop alterations in the Leydig cell compartment. These alterations range from abnormal localization and clustering to hyperplasia or tumorous formation.

Leydig cell tumors (LCTs), although uncommon in the general population, are the most frequent non-germ cell testicular neoplasms, and their incidence has been reported increasingly growing, especially in infertile patients. Given that the focal areas of Leydig cell hyperplasia are nowadays easily detectable at ultrasonography of the testis (US), as small non-palpable hypoechoic micro-nodules that can show internal vascularization, their finding create a diagnostic challenge versus low-stage malignant germ cell tumors.

Patients with testicular dysgenesis syndrome in general exhibit an elevation of Follicle-Stimulating Hormone (FSH), but in these patients, very frequently, even Luteinizing Hormone (LH) is above the reference range. The latter can work as a growth factor for Leydig cells. Since exogenous testosterone can suppress LH levels, it could be that androgen therapy could revert the LH-induced growth stimulation of Leydig cell compartment.

The purpose of this study is to evaluate the effects of androgen therapy on the size and number of non-palpable hypoechoic micro-nodules in patients with elevated gonadotropin levels.

The purpose of this study is also to evaluate whether the behavior (UltraSonographic appearance, US) of the non-palpable hypoechoic micro-nodules during a 4-month trial of testosterone therapy can offer a novel diagnostic tool in the differential diagnosis of benign versus malignant testicular nodules.

The trial will be open only for patients with multiple non-palpable hypoechoic micro-nodules that have an elevation of both FSH and LH and that are not seeking conception.

Participants in the study will be randomized to one of two treatment groups, receiving either testosterone undecanoate (low-dose androgen) or placebo, for two 6 months. All participants will be evaluated for safety at the beginning of the study and at 2, 4, and 6 months with careful history, physical examination, blood sampling and testicular ultrasonography. Patients will also be offered the possibility to perform Magnetic Resonance Imaging (MRI) of the testis at baseline and after treatment, and/or surgical enucleation of the lesions.

ELIGIBILITY:
Inclusion Criteria:

* Non-palpable Multiple hypoechoic testicular nodules (with the largest having a diameter > 2 mm and < 12 mm)
* Serum Follicle-stimulating hormone (FSH) > 7 mIU/ml (m-International-Unit/ml)
* Serum Luteinizing hormone (LH) > 7 IU (International-Unit/ml)
* Infertility: Klinefelter Syndrome, Hypergonadotropic Hypogonadism, Hypergonadotropic Azospermia, Hypergonadotropic Cryptozoospermia
* negative testicular tumors markers: beta-hCG (Human chorionic gonadotropin), alpha-FP (alpha-Feto-Protein), CEA (Carcinoembryonic antigen), LDH (Lactate dehydrogenase), ferritin, PLAP (Placental Alkaline Phosphatase).

Exclusion Criteria:

* Hypogonadotropic Hypogonadism
* FSH o LH < 7 UI
* non-homogeneous testicular lesion > 12 mm
* positive testicular tumors markers: beta-hCG, alpha-FP, CEA, LDH, ferritin, PLAP
* patients with contraindication to testosterone therapy: prostate cancer, PSA>4 ng/ml, severe hepatic or renal insufficiency, Hb>17, Htc>52%, severe urinary retention
* desire to conceive
* history of germ-cell testicular neoplasia

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2009-06; Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Nodule Size per Number | 4 month
  Percentage change of the area of the lesions multiplied by the number of the measured lesions: [(area_1 + area_2 + area_3 + ... + area_n)*n].
  The latter measure account for reduction in the number of lesions (disappearance).

SECONDARY OUTCOMES:
Nodule Size | 4 month
  Percentage change in the area of the lesion (measured with computer assisted graphics).
Luteinizing Hormone (LH) | 2 month
  Reduction of the serum Luteinizing Hormone (LH) levels during testosterone therapy
Spermatogenesis | 8 month (follow-up)
  Evaluation of sperm cell production after testosterone withdrawal.
Testicular US echo-texture | 36 month (follow-up)
  Changes in the number of areas / nodules / lesions in the long-term safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lenzi, MD, Study Chair — University of Roma La Sapienza; Andrea Isidori, MD, PhD, Principal Investigator — University of Roma La Sapienza; Vincenzo Bonifacio, MD, PhD, Study Director — University of Roma La Sapienza
Locations (1):
- Dipartimento di Fisiopatologia Medica, Rome, Lazio, Italy

REFERENCES:
- [Derived] Pozza C, Pofi R, Tenuta M, Tarsitano MG, Sbardella E, Fattorini G, Cantisani V, Lenzi A, Isidori AM, Gianfrilli D; TESTIS UNIT. Clinical presentation, management and follow-up of 83 patients with Leydig cell tumors of the testis: a prospective case-cohort study. Hum Reprod. 2019 Aug 1;34(8):1389-1403. doi: 10.1093/humrep/dez083. PMID 31532522